CLINICAL TRIAL: NCT03062163
Title: Efficacy and Safety of Resveratrol and Lipoic Acid Transdermal Patch for Lipolysis in Overweight Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: nanolab817
Record Dates: First submitted 2017-02-13; First posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Lipolysis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resveratrol lipoic Acid (Experimental): lipoic and resveratrol was loaded on the patch
  Interventions: Other: Resveratrol lipoic Acid
- Placebo (Experimental): normal saline was loaded on transdermal patch
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Resveratrol lipoic Acid — Transdermal patch loaded with resveratrol and lipoic acid
  Arms: Resveratrol lipoic Acid
Other: Placebo — Transdermal patch loaded with normal saline
  Arms: Placebo

SUMMARY:
To evaluate the lipolysis effect of resveratrol and lipoic acid transdermal patch in overweight volunteers

DETAILED DESCRIPTION:
66 participants with overweight received a resveratrol and lipoic acid transdermal patch treatment. The treatment areas have been treated including left and right arms. Subjects were evaluated using standardized measurements of body weight and circumference of arms at baseline and 2 weeks follow-up visits. Evaluation of physician were also measured.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers with BMI > 23

Exclusion Criteria:

* resveratrol or lipoic acid allergies

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2017-01-23 (Actual); Primary Completion 2017-02-06 (Actual); Study Completion 2017-02-06 (Actual)

PRIMARY OUTCOMES:
fat thickness measured | 2 weeks
  fat thickness measurement by ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Amornpun Sereemaspun, MD., Ph.D, Study Director — Chulalongkorn University
Locations (1):
- Faculty of Medicine, Chulalongkorn University, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No